CLINICAL TRIAL: NCT05381545
Title: Laser Puncture and Program of Lifestyle Modification in Lupus Females: Lipid Profile Response
Brief Title: Laser Puncture and Program of Lifestyle Modification in Lupus Females
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of Physical Therapy for Cardiovascular / Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003660
Record Dates: First submitted 2022-05-12; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): This 32-patient research group will receive, for 12 weeks, energy expenditure program (Pilates exercise, managed 5 times per week, combined with low calorie diet for).This research group will receive an additional laser puncture (with 3-time per-week design). The following points will be directly contacted by laser, for two minutes: GB34&28, ST25&36&40, SP6, and CV4&9&12.
  Interventions: Behavioral: laser puncture, energy expenditure programming, and low-calories recommended diet programming
- Group B (Active Comparator): This 32-patient research group will receive, for 12 weeks, energy expenditure program (Pilates exercise, managed 5 times per week, combined with low calorie diet ).
  Interventions: Behavioral: energy expenditure programming and low-calories recommended diet programming

INTERVENTIONS:
Behavioral: laser puncture, energy expenditure programming, and low-calories recommended diet programming — This research group will receive, for 12 weeks, energy expenditure program (Pilates exercise, managed 5 times per week) combined with low calorie diet .This research group will receive an additional laser puncture (with 3-time per-week design). The following points will be directly contacted by laser, for two minutes: GB34&28, ST25&36&40, SP6, and CV4&9&12.
  Arms: group A
Behavioral: energy expenditure programming and low-calories recommended diet programming — This research group will receive, for 12 weeks, energy expenditure program (Pilates exercise, managed 5 times per week) combined with low calorie diet.
  Arms: Group B

SUMMARY:
Serum lipid profile was significantly dysregulated in female systemic lupus erythematosus (SLE) patients

DETAILED DESCRIPTION:
the research will recruit 64 female systemic lupus erythematosus (SLE) obese patients to divide them to two study groups equally. the study groups will receive, for 12 weeks, energy expenditure program (Pilates exercise, managed 5 times per week, combined with low calorie diet for).One group only will receive an additional laser puncture (with 3-time per-week design). The following points will be directly contacted by laser, for two minutes: GB34&28, ST25&36&40, SP6, and CV4&9&12.

ELIGIBILITY:
Inclusion Criteria:

* obese female participants
* Lupus females

Exclusion Criteria:

* pregnant lupus female
* lactating lupus females
* neurologic or articular disorders
* another autoimmune conditions

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — self-representation of gender identity.
Enrollment: 64 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
triglycerides | 12 weeks
  a lipid component will be measured in blood of females

SECONDARY OUTCOMES:
high density lipoprotein | 12 weeks
  a lipid component will be measured in blood of females
cholesterol | 12 weeks
  a lipid component will be measured in blood of females
low density lipoprotein | 12 weeks
  a lipid component will be measured in blood of females

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy Cairo University, Giza, Dokki, Egypt